CLINICAL TRIAL: NCT00278278
Title: Treatment of Children and Adolescents With Diffuse Intrinsic Pontine Glioma and High Grade Glioma
Brief Title: Combination Chemotherapy and Radiation Therapy With or Without Methotrexate in Treating Young Patients With Newly Diagnosed Gliomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Responsible Party: Christoph Kramm, University Children's Hospital
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454723; GPOH-HIT-GBM-D; EU-205100
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2008-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma; untreated childhood cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood spinal cord neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Spinal Cord Neoplasms | interventions — Cisplatin; Etoposide; Ifosfamide; Lomustine; Methotrexate; Prednisone; Vincristine

ARMS (2):
- Arm I (Experimental): Patients receive high-dose methotrexate IV over 24 hours on days 1 and 15 and leucovorin calcium IV every 6 hours on days 2-3 an 16-17. Four weeks later, patients undergo external beam radiotherapy once daily, 5 days a week, for approximately 6 weeks.
  Beginning on the first day of radiotherapy, patients receive cisplatin IV over 1 hour on days 1-5, etoposide IV over 2 hours on days 1-3, and vincristine IV on days 5, 12, 19, 26, and 33. Beginning seven days prior to completion of radiotherapy, patients receive ifosfamide IV over 1 hour and cisplatin IV over 1 hour on days 1-5, etoposide IV over 2 hours on days 1-3, and vincristine IV on day 5.
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: ifosfamide; Drug: lomustine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate
- Arm II (Active Comparator): Patients undergo external beam radiotherapy once daily, 5 days a week, for approximately 6 weeks.
  Beginning on the first day of radiotherapy, patients receive cisplatin IV over 1 hour on days 1-5, etoposide IV over 2 hours on days 1-3, and vincristine IV on days 5, 12, 19, 26, and 33. Beginning seven days prior to completion of radiotherapy, patients receive ifosfamide IV over 1 hour and cisplatin IV over 1 hour on days 1-5, etoposide IV over 2 hours on days 1-3, and vincristine IV on day 5.
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: ifosfamide; Drug: lomustine; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: etoposide — Given IV
Drug: ifosfamide — Given IV
Drug: lomustine — Given IV
Drug: methotrexate — Given IV
  Arms: Arm I
Drug: prednisone — Given IV
Drug: vincristine sulfate — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether giving methotrexate together with combination chemotherapy and radiation therapy is more effective than combination chemotherapy and radiation therapy alone in treating gliomas.

PURPOSE: This randomized phase III trial is studying giving methotrexate together with combination chemotherapy and radiation therapy to see how well it works compared to combination chemotherapy and radiation therapy alone in treating young patients with newly diagnosed gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if the addition of high-dose methotrexate prior to standard treatment improves survival of patients with malignant high-grade glioma or diffuse intrinsic pontine glioma as compared to standard treatment only.

Secondary

* Determine if the addition of high-dose methotrexate, as compared to standard treatment only, improves the tumor response of these patients.
* Determine if high-dose methotrexate, compared to standard treatment only, improves the progression-free or event-free survival of these patients.
* Determine if high-dose methotrexate, as compared to standard treatment only, improves the health status (quality of life) of these patients.
* Determine if consolidation therapy improves the overall, progression-free, or event-free survival rates as compared to the historical control group.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to tumor location includes pons (yes vs no) and complete or nearly complete resection (yes vs no).

* Surgery: All patients are encouraged to undergo radical resection of the tumor to reduce intracranial pressure, remove as much tumor tissue as possible, and obtain tumor tissue for histological diagnosis. Within 14 days after surgery, patients proceed to induction chemotherapy.
* Induction therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I:

    * High-dose methotrexate with leucovorin calcium: Patients receive high-dose methotrexate IV over 24 hours on days 1 and 15 and leucovorin calcium IV every 6 hours on days 2-3 an 16-17. Patients proceed to chemoradiotherapy 4 weeks later.
    * Chemoradiotherapy (course 1): Patients undergo external beam radiotherapy once daily, 5 days a week, for approximately 6 weeks. Beginning on the first day of radiotherapy, patients receive cisplatin IV over 1 hour on days 1-5, etoposide IV over 2 hours on days 1-3, and vincristine IV on days 5, 12, 19, 26, and 33. Patients proceed to course 2 of chemoradiotherapy 7 days prior to completion of radiotherapy.
    * Chemoradiotherapy (course 2): Patients receive ifosfamide IV over 1 hour and cisplatin IV over 1 hour on days 1-5, etoposide IV over 2 hours on days 1-3, and vincristine IV on day 5. Patients proceed to consolidation chemotherapy 4 weeks later.
  * Arm II: Patients receive chemoradiotherapy courses 1 and 2 as in arm I and proceed to consolidation chemotherapy 4 weeks later.
* Consolidation chemotherapy: Patients receive vincristine IV on days 1, 8, and 15, oral lomustine once on day 2, and oral prednisone once daily on days 1-17. Treatment repeats every 6 weeks for up to 8 courses.

Quality of life is assessed 1 week after surgery, after completion of chemoradiotherapy, at 1, 4, and 13 months after completion of consolidation chemotherapy, and then annually for 3 years.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed tumors of the brain or spinal cord, meeting one of the following criteria:

  * Histologically* confirmed diagnosis of 1 of the following high-grade gliomas:

    * Glioblastoma (WHOº IV)
    * Anaplastic astrocytoma (WHOº III)
    * Gliosarcoma (WHOº III or IV)
    * Anaplastic oligo-astrocytoma NOTE: *Histological requirement may be waived for other types of brainstem glioma
  * Radiologically proven diffuse intrinsic pontine glioma
* Second malignancy or disseminate metastases or multifocal tumors are allowed if the field of irradiation is not too large

  * No diffuse metastases making craniospinal irradiation necessary

PATIENT CHARACTERISTICS:

* No cardiorespiratory insufficiency requiring medical respiration
* No low blood pressure requiring systemic catecholamines
* No severe neurological damage (e.g., coma)
* No tetraplegia without possibility to communicate
* No other poor clinical condition
* Not pregnant
* Fertile patients must use effective contraception
* No hypersensitivity to methotrexate, cisplatin, vincristine, lomustine, or ifosfamide
* No other malignancy preceding radiotherapy that does not allow further radiation

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for brain tumor
* The following prior therapies are allowed:

  * Mistletoe
  * H15 (extract of Boswellia serrata)
  * Homeopathy therapy with dilution > 4D
  * Alternative medicine without proven efficacy
* No prior radiotherapy for brain tumor
* No concurrent alcohol or tobacco consumption
* No concurrent participation in another study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-09; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) rate at 5.5 years

SECONDARY OUTCOMES:
Comparison of OS, progression-free survival, and event-free survival with historical control annually
Long-term sequelae annually
Tumor response
Progression-free survival
Event-free survival
Health status

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kramm, MD, Study Chair — University Children's Hospital
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- [Result] Wolff JE, Kortmann RD, Wolff B, Pietsch T, Peters O, Schmid HJ, Rutkowski S, Warmuth-Metz M, Kramm C. High dose methotrexate for pediatric high grade glioma: results of the HIT-GBM-D pilot study. J Neurooncol. 2011 May;102(3):433-42. doi: 10.1007/s11060-010-0334-2. Epub 2010 Aug 8. PMID 20694800